CLINICAL TRIAL: NCT06676137
Title: China Coronary Microvascular Disease(CCMD) Registry
Brief Title: An Observational Study of Coronary Microvascular Disease of China
Acronym: CCMD
Status: Recruiting | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE202410
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood, saliva, stool and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-obstructive coronary heart disease refers to patients with angina pectoris without significant narrowing of the epicardial vessels. Coronary microvascular disease(CMD) is a kind of non-obstructive coronary heart disease, and its clinical detection rate is increasing, seriously affecting the quality of life of patients, and increasing the risk of cardiovascular adverse events, but its mechanism has not been fully understood. This study will prospectively collect patients who meet the diagnosis of CMD, observe the development and outcome of the disease, and explore its occurrence and development mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Angina symptoms
2. Objective evidence of myocardial ischemia
3. Coronary angiography was normal,irregular tube wall, or stenosis <50%

Exclusion Criteria:

1. People under the age of 18
2. Non-cardiogenic chest pain and other heart conditions such as variant angina, cardiomyopathy, myocarditis or valvular heart disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient had obvious symptoms of angina pectoris, but coronary angiography showed no obvious epicardial stenosis, and auxiliary examinations such as ultrasound, CTP,CMR, PET, SPECT, and coronary function examination indicate the presence of microcirculation dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-10-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Establish a Registry of CMD patients in China | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: muwei li, Ph.D, Study Chair — Fuwai central China cardiovascular hospotial
Locations (1):
- Fuwai central China cardiovascular hospotial, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No